CLINICAL TRIAL: NCT02432495
Title: Anterior Screw Fixation Versus Halo Immobilization of Type II Odontoid Fractures in Geriatric Patients With Increased Anesthesia Risk
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 2008/10
Record Dates: First submitted 2015-04-20; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Spinal Fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Anterior screw fixation: Patients aged 65 years or older with an ASA score of 2 or higher who had undergone anterior screw fixation of type II odontoid fractures
  Interventions: Other: ANTERIOR SCREW FIXATION
- Halo immobilization: Patients aged 65 years or older with an ASA score of 2 or higher who had undergone of halo immobilization of type II odontoid fractures
  Interventions: Other: HALOV VEST IMMOBILIZATION

INTERVENTIONS:
Other: ANTERIOR SCREW FIXATION — Patients aged 65 years or older with an ASA score of 2 or higher who had undergone anterior screw fixation of type II odontoid fractures
  Groups: Anterior screw fixation
Other: HALOV VEST IMMOBILIZATION — Patients aged 65 years or older with an ASA score of 2 or higher who had undergone halo immobilization of type II odontoid fractures
  Groups: Halo immobilization

SUMMARY:
The management of type II odontoid fractures in geriatric trauma victims remains a source of substantial controversy. The purpose of this study was to compare anterior screw fixation with halo-vest-immobilization in patients with type II odontoid fractures.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years or older with an ASA (= American society of anesthesiologists) score of 2 or higher
* complete sets of collected data and a follow-up monitoring of at least five years

Exclusion Criteria:

* type III odontoid fractures
* patients with incomplete data sets
* patients with penetrating mechanism of injury or congenital cervical spine anomalies

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: patients aged 65 years or older with an ASA score of 2 or higher who had undergone either anterior screw fixation or halo immobilization of type II odontoid fractures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
neurological deficits | at least 60 months follow up
  Neurologic deficits measured including the CSOQ (Cervical Spine Outcome Questionnaire) before and after surgery as well as compared in both procedure groups
radiographic outcome (documentation of boney union) | at least 60 months follow up
  documentation of boney union compared in both procedure groups